CLINICAL TRIAL: NCT06418503
Title: Effects of EMG-Biofeedback Balance Training on Hoffman's Reflex and Their Longevity
Brief Title: Effects of EMG-Biofeedback Balance Training on Hoffman's Reflex
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17485
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Spinal Reflex Excitability; Balance
Keywords: Hoffman's; Reflex; Biofeedback; EMG

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be masked to which intervention they receive (balance training or EMG-biofeedback balance training).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance Training (Sham Comparator): Completing a Tetris (block stacking) computer game while attached to an EMG device by electrodes and leads.
  Interventions: Other: Balance Training
- EMG-Biofeedback Training (Experimental): Completing an EMG-biofeedback block stacking game using the electrodes to detect muscle signals which are controlling the movements of the blocks.
  Interventions: Other: EMG-Biofeedback Training

INTERVENTIONS:
Other: Balance Training — Participants will complete 16 sessions of balance training (30 min. each) over one month.
  Arms: Balance Training
Other: EMG-Biofeedback Training — Participants will complete 16 sessions of EMG-biofeedback balance training (30 min. each) over one month.
  Arms: EMG-Biofeedback Training

SUMMARY:
The purpose of this study is to gain a further understanding of the effects of EMG-biofeedback balance training and we will be analyzing changes in spinal reflex excitability by responses from the calve muscles and data about your standing balance. The EMG-biofeedback balance training has the potential to improve balance of older adults and prevent future falls and in this study we will learn if it also creates changes in the nervous system.

This study aims to 1) determine the effects of a one-month long EMG-biofeedback balance intervention on the H-reflex amplitude, 2) determine whether there is a related behavioural change in the control of balance and 3) determine whether changes in balance and H-reflex amplitude persist for up to two weeks following the end of the balance training intervention.

DETAILED DESCRIPTION:
Injuries caused by falls are a major worldwide issue and the most serious injuries include hip fractures and trauma to the brain. In-depth analysis of the risk factors for falls have discovered that balance disorders and abnormal gait are the strongest contributors. It is not a surprise that neural control of posture is altered as a function of age. Falls among the elderly has become an increasing issue and are leading to an escalating number of medical conditions, mortality and utilization of health care services. In Canada, 32 to 42% of older adults who are 70 years or older fall each year. Balance is the key ability needed to avoid falls because maintaining upright balance is needed to complete individual daily activities. Quantitative assessments are needed when evaluating the postural balance of participants. The force plate is a piece of equipment that is a reliable balance assessment method which is used widely in both laboratory and clinical settings. Despite the many research studies over the last three decades analyzing the effects of age and postural control, the number of deaths caused by falling and fall-related injuries has continued to increase. More studies are needed to highlight how old age affects neural mechanisms of postural control. Specifically, we need to understand the mechanisms by which balance training can lead to improved postural control to decrease falls among older adults.

A valuable neurophysiological measurement known as the Hoffman (H) reflex, has a high sensitivity to posture. Measuring the H-reflex amplitude can be used to detect whether changes in spinal excitability accompany balance training. It is a relatively simple technique which makes it an intriguing tool for research. The H-reflex has been used for decades in motor control studies which emphasize spinal mechanisms. It is commonly used as a tool for analyzing spinal excitability, or how effectively synaptic transmission occurs between motor neurons and 1a afferents.

For balance training, electromyography (EMG) biofeedback can be implemented which would involve the participants controlling objects on a screen through the electrical signals of their muscles while standing. The sensors used for EMG are not painful or invasive and can be applied to target the impairment of specific muscles or muscle groups. The EMG-Biofeedback system creates a classifier that predicts the user's intended game control inputs through real-time EMG signals. This innovation would be achieved by placing the sensors on the upper leg and arms to collect data for the signals of the lower and upper extremities, so the motor performance and successful game execution can be focused on the balance of participants. Eighteen sessions (40 minutes each) of EMG-biofeedback training of the lower body (tibialis anterior muscle) over three weeks in participants suffering with chronic stroke was shown to improve motor control outcomes including balance and strength.

To gain a further understanding of the neurophysiological effects of EMG-biofeedback, we will be analyzing changes in spinal reflex excitability by measuring H-reflex amplitudes, and balance board test results before and after 4 weeks of balance training in the aging population. While there have been published studies regarding this intervention improving balance, there have not been any studies exploring whether EMG-biofeedback training also changes spinal reflex excitability. This intervention has the potential to improve spinal reflexes and balance of older adults and prevent future falls. This intervention can possibly decrease major injuries across the healthy older adult population, and changes in H-reflex amplitudes can be associated with balance changes. Studies which have explored changes in H-reflex amplitude after one-month long balance training, have not done a follow-up assessment to confirm the longevity of improvements in balance and decreased amplitudes of the H-reflex.

Methods:

During the participants' first visit to the laboratory, they will complete 3 functional assessments, and one neurophysiological assessment. The functional assessments will measure balance in a standing position. These balance assessments will take approximately 10 min. to complete. The measurement of muscle activity will involve non-invasive stimulation behind the knee which will evoke a muscle twitch in the calve (soleus) muscle. This Hoffman Reflex assessment will be completed for each leg and reflects the activity of circuits within the spinal cord that are thought to contribute to balance. This procedure requires approximately 20 minutes for each leg.

The participants will be randomly assigned to the balance training or biofeedback balance training group by the lead investigator of this study, and the participant will not be told which group they have been assigned to. Irrespective of which group the participant has been assigned to, they will have electrodes placed on upper and lower body muscles which will be attached to the EMG system using leads and you will be completing a computer game that requires your balance for 30 min. each of your training sessions. Assistive devices such as canes, walkers etc. will not be used during the balance training. The participants can take breaks and sit down occasionally during the balance training. This training will take place 4 times per week for a total of 16 times. Both groups will experience the computer game during standing balance training.

The day after their last session, they will complete a follow-up assessment session which will also involve completion of the 3 functional balance tests and measurement of muscle activity for each leg, which will follow the same procedure as the first assessment session.

The second follow-up assessment will take place 2 weeks after the final training session. All assessments from the first follow-up will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy older adults between 60-75 years old
* able to stand free of assistive devices for at least 3 consecutive minutes
* free of visual disorders that prevent meaningful interaction with the intervention interface.

Exclusion Criteria:

* Sustained a serious musculoskeletal injury in the past 6 months or have any diagnosis that could impact movement coordination or balance
* significant cognitive or language barriers

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in Spinal Reflex Excitability | Pre-intervention (before 1st training session), post-intervention (1-2 days after last training session), 2-week follow-up
  Measurements of maximal Hoffman reflex
Change in Balance | Pre-intervention (before 1st training session), post-intervention (1-2 days after last training session), 2-week follow-up
  Measurements of balance using balance board assessments

REFERENCES:
- [Background] Chen B, Liu P, Xiao F, Liu Z, Wang Y. Review of the Upright Balance Assessment Based on the Force Plate. Int J Environ Res Public Health. 2021 Mar 8;18(5):2696. doi: 10.3390/ijerph18052696. PMID 33800119
- [Background] Bakker LBM, Lamoth CJC, Vetrovsky T, Gruber M, Caljouw SR, Nieboer W, Taube W, van Dieen JH, Granacher U, Hortobagyi T. Neural Correlates of Balance Skill Learning in Young and Older Individuals: A Systematic Review and Meta-analysis. Sports Med Open. 2024 Jan 7;10(1):3. doi: 10.1186/s40798-023-00668-3. PMID 38185708
- [Background] Tsaih PL, Chiu MJ, Luh JJ, Yang YR, Lin JJ, Hu MH. Practice Variability Combined with Task-Oriented Electromyographic Biofeedback Enhances Strength and Balance in People with Chronic Stroke. Behav Neurol. 2018 Nov 26;2018:7080218. doi: 10.1155/2018/7080218. eCollection 2018. PMID 30598705
- [Background] Theodosiadou A, Henry M, Duchateau J, Baudry S. Revisiting the use of Hoffmann reflex in motor control research on humans. Eur J Appl Physiol. 2023 Apr;123(4):695-710. doi: 10.1007/s00421-022-05119-7. Epub 2022 Dec 26. PMID 36571622
- [Background] Park C, Mishra RK, York MK, Enriquez A, Lindsay A, Barchard G, Vaziri A, Najafi B. Tele-Medicine Based and Self-Administered Interactive Exercise Program (Tele-Exergame) to Improve Cognition in Older Adults with Mild Cognitive Impairment or Dementia: A Feasibility, Acceptability, and Proof-of-Concept Study. Int J Environ Res Public Health. 2022 Dec 6;19(23):16361. doi: 10.3390/ijerph192316361. PMID 36498431
- [Background] Public Health Agency of Canada. (2022). Senior-falls-in-Canada-en.pdf. Surveillance Report on Falls Among Older Adults in Canada. https://www.canada.ca/content/dam/hc-sc/documents/reserch/surveillance/senior-falls-in-Canada-en.pdf